CLINICAL TRIAL: NCT00807365
Title: Six Month Treatment of GHRH in the Elderly
Brief Title: Six Month Treatment of Growth Hormone Releasing Hormone (GHRH) in the Elderly
Acronym: PP2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left JHU
Sponsor: Johns Hopkins University (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00005793; 2002P-001781; P01-AG0059-21
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Results first posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-03

CONDITIONS: Elderly
Keywords: Growth Hormone-Releasing Hormone; Growth Hormone Insufficiency; Aging; Growth Hormone; Physiological Effects of Drugs; Hormones, Hormone Substitutes, and Hormone Antagonists; Hormones
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Growth Hormone-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GHRH (Experimental): Growth Hormone-Releasing Hormone
  Interventions: Drug: GHRH

INTERVENTIONS:
Drug: GHRH — GHRH administered subcutaneously at 2.0 mg/kg/dose bolus each night at 11:00 Post Meridian (PM), 1:00 Ante Meridian (AM), 3:00 AM, & 5:00 AM for 6 months.
  Other Names: Growth Hormone-Releasing Hormone

SUMMARY:
The purpose of the study is to evaluate the effect of a naturally occurring hormone, called Growth Hormone Releasing Hormone (GHRH), on the muscle, bone and fat tissues of the body. GHRH stimulates the production of growth hormone (GH), which regulates the build up of many tissues in the body, including muscles and bones. Many elderly people have low levels of GH. The overall goal of this research is to determine the effectiveness of GHRH to raise levels of GH and improve these body tissues. The purpose of the tests is to measure how the body handles sugar, fat, and proteins. GH can affect your body's use of sugar, fat and proteins.

DETAILED DESCRIPTION:
Growth hormone (GH) is a major anabolic hormone that exerts important stimulatory effects on protein synthesis. Many of the peripheral tissue effects of GH are mediated by insulin-like growth factor I (IGF-I), produced systemically by the liver or locally in tissues in response to GH stimulation. IGF-I in turn regulates GH secretion by negative feedback mechanisms at the pituitary gland. Several investigators have shown that aging is associated with a decrease in spontaneous GH secretion and IGF-I levels. GH levels decline by 14% for each decade after puberty, and, in healthy 59-98 year old men, IGF-I levels below the 2.5 percentile of younger men are present in 85%. Reduction of GH release in aging is thought to be associated with an increase in somatostatin tone, decrease in hypothalamic GHRH output, and diminished response to GHRH. The fact that aging is accompanied by a decrease in protein synthesis leading to a loss of lean body mass (LBM) and a gain in body fat suggests that a decrease in GH secretion may contribute to these changes. It has been hypothesized that restoration of GH level in the elderly to the levels observed in younger individuals may lead to improvements in body composition.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of low GH levels as assessed by a fasting IGF-1 level <135ng/ml.
* Volunteers whose BMI is above normal range and below extreme obesity (BMI 25-40 kg/m2).

Exclusion Criteria:

* Diabetes.
* Known coronary artery disease.
* Liver, peptic or inflammatory bowel disease. Renal or hematologic disease.
* Hematocrit <30% or >50%.
* Clinically significant prostate hypertrophy.
* Elevated Prostate specific antigen (PSA) (4ng/ml).
* Prostate & breast cancer.
* History of malignancy <5 years other than basal cell of the skin.
* Chronic pulmonary disease or other systemic disorders.
* Use of certain drugs (such as thiazide diuretics, beta-blockers, steroids (except for replacement doses), coumadin, and or androgen supplements).
* Peanut allergy.
* Gross physical impairment.
* Sleep apnea.
* Uncontrolled hypertension(blood pressure >160/95 and or requiring more than two antihypertensive medications).
* A clinically worrisome mammogram in women.
* Exercise training (>2x/wk for 20 min at a level that produces sweating) in the last 6 months.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-12-17 (Actual); Primary Completion 2010-04-29 (Actual); Study Completion 2010-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dariush Elahi, PhD, Principal Investigator — Johns Hopkins University; Kenneth L. Minaker, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GHRH
Started | 5
Completed | 0
Not Completed | 5
Not completed — Study Terminated | 5

BASELINE CHARACTERISTICS:
Groups:
- GHRH: Growth Hormone-Releasing Hormone
  GHRH: GHRH administered subcutaneously at 2.0 mg/kg/dose bolus each night at 11:00 PM, 1:00 AM, 3:00 AM, & 5:00 AM for 6 months.
Arm/Group | GHRH
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Lean Body Mas
Time Frame: 2 years
Population: Study terminated prior to collection of data
Arm/Group | GHRH
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | GHRH
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes